CLINICAL TRIAL: NCT07372664
Title: External Validation of the Volume-Velocity Index for Weaning Prediction: a Multicenter Observational Study
Brief Title: External Validation of VVI
Acronym: E-VVI
Status: Recruiting | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, DEMOSTHENES MAKRIS, Professor of Intensive Care, Director of the Department of Intensive Care, General University Hospital of Larissa, University of Thessaly
Other Study IDs: 23/17/16-12-25
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Weaning Mechanical Ventilation
Keywords: weaning; mechanical ventilation; ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing weaning

SUMMARY:
Failure of liberation from mechanical ventilation increases days spent being mechanically ventilated, the length of stay and the morbidity of patients. Thus it is crucial that those patients who are ready to be liberated are accurately detected. In this study the investigators want to externally validate an index (the volume-velocity index, VVI) which in a preliminary study was found to predict with high accuracy the outcome of ventilator liberation.

In this study, in patients who are deemed ready to undergo weaning by their treating physician the investigators will measure the excursion of the diaphragm, the principal respiratory muscle, the inspiratory time and the tidal volume and the volume breathed by the patient at each respiration in three phases:

1. during pressure support ventilation with 5/5,
2. during pressure support ventilation with 8/0,
3. during t-tube or pressure support ventilation with 0/0. All of these phases are ventilatory modalities widely used during weaning from mechanical ventilation.

The investigators will evaluate whether VVI can predict accurately the weaning outcome.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients for more than 48h
* First Spontaneous breathing trial
* Deemed as ready to undergo weaning by the treating physician, according to published readiness criteria (DOI: 10.1183/09031936.00010206)

Exclusion Criteria:

* pregnant patients
* preexisting diaphragmatic disease or injury
* tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical Care patients undergoing weaning from mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Weaning outcome | From the start of the spontaneous breathing trial to failure or success at 48 hours after exubation.
  Validate the predictive capability of VVI for weaning outcome

SECONDARY OUTCOMES:
VVI for SBT or extubation | From the start of the spontaneous breathing trial to failure or success at 48 hours after exubation.
  Comparison of the capability of VVI to predict SBT or extubation failure

OTHER OUTCOMES:
VVI vs RSBI | From the start of the spontaneous breathing trial to failure or success at 48 hours after exubation.
  Comparison of the predictive capability of VVI with RSBI for weaning outcome
Predictive capability of VVI between long or short ventilation time | From the start of the spontaneous breathing trial to failure or success at 48 hours after exubation.
  Comparison of the redictive capability of VVI between patients ventilated for more than 7 days with patients ventilated for less than 7 days
VVI in various SBT modalities | From the start of the spontaneous breathing trial to failure or success at 48 hours after exubation.
  Compare the ability of VVI to predict the weaning outcome in various SBT modalities, namely Pressure Support 8/0 and Pressure Support 5/5 versus t-tube or Pressure Support 0/0
Relationship of VVI with MIP and MRC | From the start of the spontaneous breathing trial to failure or success at 48 hours after exubation.
  evaluate the relationship of VVI with indices of strength status such as the maximal inspiratory pressure, for the respiratory muscles, and the medical research council score, for the ICU acquired weakness.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos - Alkiviadis Menis, Principal Investigator — General university hospital of larissa; Demosthenes Makris, Study Director — University of Thessaly
Locations (3):
- Greece (3):
  - General University Hospital of Larissa, Larissa
  - AHEPA - University General Hospital, Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki

IPD SHARING:
Plan to Share IPD: No